CLINICAL TRIAL: NCT02729883
Title: A Pilot Study of 'Take the Fight' as Community-Based Participatory Research
Brief Title: Take the Fight in Supporting and Empowering Patients With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Issue
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00037093; NCI-2016-00384 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99216 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Healthy Subject; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (Take the Fight) (Experimental): Patients receive patient navigation via strategists from the Take the Fight for 8 weeks. Patients also complete interviews regarding perceived physical, logistical, psychosocial, and informational challenges experienced prior to meeting with strategists/navigators and how challenges were addressed by navigator or others, perceived benefits or limitations of navigator assistance. Strategists also complete interviews regarding their perceptions on how patients benefited from participation, challenges patients experienced that were directly or indirectly related to their cancer diagnosis and treatment, how these concerns were addressed, barriers to addressing these concerns, and patient health literacy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Supportive Care

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete interviews
Procedure: Supportive Care — Receive patient navigation via the Take the Fight strategists
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This pilot clinical trial studies Take the Fight in supporting and empowering patients with cancer through their treatment process. Patients with cancer are faced with many obstacles created by the current state of the healthcare system. The purpose of Take the Fight is to train college students, also called patients' navigators or strategists, to assist and support patients to navigate into the healthcare system and receive the care they need. The strategists are matched with patients and attend/coordinate most patients' medical appointments. The strategists also advance communications between the patient and the medical staff to facilitate both the exchange of medical information as well as increase the patient's compliance with treatment. Take the Fight may improve the health and quality of life outcomes of cancer patients during critical treatment periods by increasing treatment compliance, eliminating barriers to better care, and increasing clinical trial participation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Delineate the benefits of and limitations to having Take the Fight strategists, performing as lay-navigators, as perceived by both the patients and the students.

SECONDARY OBJECTIVES:

I. Investigate changes in self-reported outcomes for patients and the Take the Fight strategists.

OUTLINE:

Patients receive patient navigation via strategists from the Take the Fight for 8 weeks. Patients also complete interviews regarding perceived physical, logistical, psychosocial, and informational challenges experienced prior to meeting with strategists/navigators and how challenges were addressed by navigator or others, perceived benefits or limitations of navigator assistance. Strategists also complete interviews regarding their perceptions on how patients benefited from participation, challenges patients experienced that were directly or indirectly related to their cancer diagnosis and treatment, how these concerns were addressed, barriers to addressing these concerns, and patient health literacy.

After completion of study, patients and strategists are followed up for 8-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS ELIGIBILITY CRITERIA
* Have histologically confirmed cancer
* Karnofsky performance scale (KPS) score of >= 60
* The ability to understand and be willing to sign an informed consent document
* Willing to undergo a form of cancer therapy and subsequent follow-up care
* STRATEGISTS INCLUSION CRITERIA
* Age >= 18 years
* Wake Forest University student
* Have volunteered as a student strategist at Comprehensive Cancer Center of Wake Forest University (CCCWFU); all strategists are required to have gone through Take the Fight (TTF) training prior to their volunteer work

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in patients self-reported outcomes using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life-Cancer 30 (QLQ-C30) questionnaire | Baseline to up to 18 weeks
  Descriptive statistics will be measured, including frequencies, percentages, means and standard deviations of patient self-report measures will be calculated. Ninety-five percent confidence intervals will also be calculated for the outcomes measures at each time point.
Change in strategists self-reported outcomes using Caregiver Quality of Life Index-Cancer (CQOLC, McMillian, 1996) scale | Baseline to up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grant, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States